CLINICAL TRIAL: NCT00891202
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study Confirming the Efficacy and Safety of Genz-112638 in Patients With Gaucher Disease Type 1 (ENGAGE)
Brief Title: A Study of Eliglustat Tartrate (Genz-112638) in Patients With Gaucher Disease (ENGAGE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GZGD02507; 2008-005222-37 (EudraCT Number); EFC12813 (Other: Sanofi)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Gaucher Disease, Type 1
Keywords: Gaucher,; beta-glucosidase,; acid ß-glucosidase,; glucocerebrosidase,; glucosylceramide,; D-glucosyl-N-acylsphingosine glucohydrolase,; substrate reduction therapy
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Eliglustat
  Interventions: Drug: Eliglustat tartrate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eliglustat tartrate — PAP: Eliglustat tartrate (ET) capsule 50 mg orally on Day 1 followed by ET 50 mg capsule twice daily (BID) from Day 2 to Week 4, then either ET 50 mg capsule BID (participants with Genz-99067 [active moiety of ET in plasma] trough plasma concentration >=5 ng/mL) or ET 100 mg capsule BID (participants with Genz-99067 trough plasma concentration <5 ng/mL), up to Week 39. PK assessment at Week 2 used for dose adjustment after Week 4. LTTP: Participants of the eliglustat arm in PAP who completed PAP were included in LTTP and received ET capsule 50 mg BID orally from Day 1 (post Week 39) until Week 43 followed by ET 50 mg or 100 mg capsule BID up to Week 47, then ET 50 mg or 100 mg or 150 mg capsule BID up to Week 312. Dose adjustments at Week 43 and Week 47 were based on Genz-99067 trough plasma concentrations (if trough plasma concentration <5 ng/mL: next higher dose administered; if >=5 ng/mL: same dose continued) at Week 41 & Week 45, respectively.
  Other Names: Genz-112638
  Arms: Active
Drug: Placebo — PAP: Matching placebo capsule once daily on Day 1 followed by matching placebo capsule BID from Day 2 through Week 39. LTTP: Participants of the placebo arm in PAP who completed PAP were included in LTTP and received eliglustat tartrate from Day 1 (post Week 39) up to Week 312. Day 1 (post Week 39) was considered as baseline for LTTP. On Day 1, participants received eliglustat tartrate capsule 50 mg BID orally until Week 43 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 47, then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to Week 312. Dose adjustments at Week 43 and Week 47 were based on Genz-99067 trough plasma concentrations (if trough plasma concentration <5 ng/mL: next higher dose administered; if >=5 ng/mL: same dose continued) at Week 41 & Week 45, respectively.
  Arms: Placebo

SUMMARY:
This Phase 3 study was designed to confirm the efficacy and safety of eliglustat tartrate (Genz-112638) in participants with Gaucher disease Type 1.

DETAILED DESCRIPTION:
Gaucher disease is characterized by lysosomal accumulation of glucosylceramide due to impaired glucosylceramide hydrolysis. Type 1 Gaucher disease, the most common form accounts for greater than (>) 90% of cases and does not involve the central nervous system (CNS). Typical manifestations of Type 1 Gaucher disease include splenomegaly, hepatomegaly, thrombocytopenia, anemia, skeletal pathology and decreased quality of life. The disease manifestations are caused by the accumulations of glucosylceramide (storage material) in Gaucher cells which have infiltrated the spleen and liver as well as other tissue. Eliglustat tartrate is a small molecule developed as an oral therapy which acts to specifically inhibit production of this storage material in Gaucher cells.

This study was designed to determine the efficacy, safety, and pharmacokinetics (PK) of eliglustat tartrate in adult participants (>16 years) with Gaucher disease Type 1. The study consisted of 2 periods: The Double-Blind Primary Analysis Period (PAP [Day 1 to Week 39]) and the Long Term Treatment Period (LTTP/Open-Label Period (post-Week 39 [Day 1 of the Open-Label Period] through study completion).

ELIGIBILITY:
Inclusion Criteria:

* The participant (and/or their parent/legal guardian) was willing and able to provide signed informed consent prior to any study-related procedures to be performed;
* The participant was at least 16 years old at the time of randomization;
* The participant had a confirmed diagnosis of Gaucher disease Type 1;
* Female participants of childbearing potential must had a documented negative pregnancy test prior to dosing. In addition all female participants of childbearing potential must use a medically accepted form of contraception throughout the study.

Exclusion Criteria:

* The participant has had a partial or total splenectomy;
* The participant had received pharmacological chaperones or miglustat within 6 months prior to randomization;
* The participant had received enzyme replacement therapy within 9 months prior to randomization;
* The participant had Type 2 or 3 Gaucher disease or was suspected of having Type 3 Gaucher disease;
* The participant had any clinically significant disease, other than Gaucher disease, including cardiovascular, renal, hepatic, gastrointestinal (GI), pulmonary, neurologic, endocrine, metabolic, (for example, hypokalemia, hypomagnesemia), or psychiatric disease, other medical conditions, or serious intercurrent illness that might confound the study results, or, on the opinion of the investigator, might preclude participation in the study;
* The participant had tested positive for the human immunodeficiency virus (HIV) antibody, Hepatitis C antibody, or Hepatitis B surface antigen;
* The participant had received an investigational product within 30 days prior to randomization;
* The participant was pregnant or lactating.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (18):
- United States (6):
  - UCSF MS Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University Medical Genetics, Decatur, Georgia
  - University of Kansas Medical Center, Division of Hematology/Oncology, Dept. of Medicine, Westwood, Kansas
  - New York University School of Medicine, Neurology Department, New York, New York
  - Mount Sinai School of Medicine, New York, New York
- University hospital "Alexandrovska" Sofia, Sofia, Bulgaria
- Canada (2):
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
  - Mount Sinai Hospital and the Samuel Lunenfeld Research Institute, Toronto Ontario
- Hospital de San Jose, Bogotá, Colombia
- Christian Medical College Hospital, Vellore, India
- Rabin Medical Center, Beilinson Hospital, Petach Tikvah, Israel
- Hôtel-Dieu de France University Hospital, Beirut, Lebanon
- OCA Hospital, Monterrey, Nuevo Leon, Mexico
- Hematology Research Center of Ministry of Healthcare of the Russian Federation, Moscow, Russia
- Institut za endokrinologiju, Belgrade, Serbia
- Hopital La-Rabta, Tunis, TN, Tunisia
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Background] Lukina E, Watman N, Arreguin EA, Banikazemi M, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Rosenthal DI, Kaper M, Singh T, Puga AC, Bonate PL, Peterschmitt MJ. A phase 2 study of eliglustat tartrate (Genz-112638), an oral substrate reduction therapy for Gaucher disease type 1. Blood. 2010 Aug 12;116(6):893-9. doi: 10.1182/blood-2010-03-273151. Epub 2010 May 3. PMID 20439622
- [Background] Lukina E, Watman N, Arreguin EA, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Kamath RS, Rosenthal DI, Kaper M, Singh T, Puga AC, Peterschmitt MJ. Improvement in hematological, visceral, and skeletal manifestations of Gaucher disease type 1 with oral eliglustat tartrate (Genz-112638) treatment: 2-year results of a phase 2 study. Blood. 2010 Nov 18;116(20):4095-8. doi: 10.1182/blood-2010-06-293902. Epub 2010 Aug 16. PMID 20713962
- [Background] McEachern KA, Fung J, Komarnitsky S, Siegel CS, Chuang WL, Hutto E, Shayman JA, Grabowski GA, Aerts JM, Cheng SH, Copeland DP, Marshall J. A specific and potent inhibitor of glucosylceramide synthase for substrate inhibition therapy of Gaucher disease. Mol Genet Metab. 2007 Jul;91(3):259-67. doi: 10.1016/j.ymgme.2007.04.001. Epub 2007 May 16. PMID 17509920
- [Background] Peterschmitt MJ, Burke A, Blankstein L, Smith SE, Puga AC, Kramer WG, Harris JA, Mathews D, Bonate PL. Safety, tolerability, and pharmacokinetics of eliglustat tartrate (Genz-112638) after single doses, multiple doses, and food in healthy volunteers. J Clin Pharmacol. 2011 May;51(5):695-705. doi: 10.1177/0091270010372387. Epub 2010 Sep 23. PMID 20864621
- [Background] Kamath RS, Lukina E, Watman N, Dragosky M, Pastores GM, Arreguin EA, Rosenbaum H, Zimran A, Aguzzi R, Puga AC, Norfleet AM, Peterschmitt MJ, Rosenthal DI. Skeletal improvement in patients with Gaucher disease type 1: a phase 2 trial of oral eliglustat. Skeletal Radiol. 2014 Oct;43(10):1353-60. doi: 10.1007/s00256-014-1891-9. Epub 2014 May 10. PMID 24816856
- [Background] Lukina E, Watman N, Dragosky M, Pastores GM, Arreguin EA, Rosenbaum H, Zimran A, Angell J, Ross L, Puga AC, Peterschmitt JM. Eliglustat, an investigational oral therapy for Gaucher disease type 1: Phase 2 trial results after 4 years of treatment. Blood Cells Mol Dis. 2014 Dec;53(4):274-6. doi: 10.1016/j.bcmd.2014.04.002. Epub 2014 May 15. PMID 24835462
- [Result] Mistry PK, Lukina E, Ben Turkia H, Amato D, Baris H, Dasouki M, Ghosn M, Mehta A, Packman S, Pastores G, Petakov M, Assouline S, Balwani M, Danda S, Hadjiev E, Ortega A, Shankar S, Solano MH, Ross L, Angell J, Peterschmitt MJ. Effect of oral eliglustat on splenomegaly in patients with Gaucher disease type 1: the ENGAGE randomized clinical trial. JAMA. 2015 Feb 17;313(7):695-706. doi: 10.1001/jama.2015.459. PMID 25688781
- [Derived] Peterschmitt MJ, Foster MC, Ji AJ, Zajdel MB, Cox GF. Plasma glucosylsphingosine correlations with baseline disease burden and response to eliglustat in two clinical trials of previously untreated adults with Gaucher disease type 1. Mol Genet Metab. 2023 Mar;138(3):107527. doi: 10.1016/j.ymgme.2023.107527. Epub 2023 Jan 25. PMID 36739645
- [Derived] Mistry PK, Lukina E, Ben Turkia H, Shankar SP, Baris Feldman H, Ghosn M, Mehta A, Packman S, Lau H, Petakov M, Assouline S, Balwani M, Danda S, Hadjiev E, Ortega A, Foster MC, Gaemers SJM, Peterschmitt MJ. Clinical outcomes after 4.5 years of eliglustat therapy for Gaucher disease type 1: Phase 3 ENGAGE trial final results. Am J Hematol. 2021 Sep 1;96(9):1156-1165. doi: 10.1002/ajh.26276. Epub 2021 Jul 11. PMID 34161616

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 72 participants were screened between 5 November 2009 and 29 July 2011, of which 32 participants were screen failure. Overall 40 participants were enrolled and the study was conducted across 18 centers in 12 countries.
Pre-assignment Details: The 40 participants who met inclusion criteria received placebo or Genz-112638 (eliglustat tartrate) during 39 weeks primary analysis period (PAP). After Week 39 of the PAP, all participants who remained in the study received eliglustat tartrate in the long-term treatment period (LTTP) for up to Week 312.
Groups:
- PAP: Eliglustat: Eliglustat tartrate capsule as a single 50 milligram (mg) dose on Day 1 followed by eliglustat tartrate 50 mg capsule twice daily (BID) from Day 2 to Week 4, and then either eliglustat tartrate 50 mg capsule BID (in participants who had a Genz-99067 [active moiety of eliglustat tartrate in plasma] trough plasma concentration greater than or equal to [>=] 5 nanogram per milliliter [ng/mL]) or eliglustat tartrate 100 mg capsule BID (in participants who had a Genz-99067 trough plasma concentration less than [<] 5 ng/mL), up to Week 39. The pharmacokinetic (PK) assessment at Week 2 was used for dose adjustment after Week 4.
- PAP: Placebo: Matching placebo capsule once daily on Day 1 followed by matching placebo capsule BID from Day 2 through Week 39.
- LTTP: Eliglustat (Originally on Eliglustat): Participants of the eliglustat arm in PAP who completed PAP were included in LTTP and received eliglustat tartrate capsule 50 mg BID orally from Day 1 (post Week 39) until Week 43 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 47, then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to Week 312. Dose adjustments at Week 43 and Week 47 were based on Genz-99067 trough plasma concentrations (if trough plasma concentration <5 ng/mL: next higher dose administered; if >=5 ng/mL: same dose continued) at Week 41 & Week 45, respectively.
- LTTP: Eliglustat (Originally on Placebo): Participants of the placebo arm in PAP who completed PAP were included in LTTP and received eliglustat tartrate from Day 1 (post Week 39) up to Week 312. Day 1 (post Week 39) was considered as baseline of LTTP for this arm. On Day 1, participants received eliglustat tartrate capsule 50 mg BID orally until Week 43 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 47, then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to Week 312. Dose adjustments at Week 43 and Week 47 were based on Genz-99067 trough plasma concentrations (if trough plasma concentration <5 ng/mL: next higher dose administered; if >=5 ng/mL: same dose continued) at Week 41 & Week 45, respectively.
Period: PAP (Up To Week 39)
Arm/Group | PAP: Eliglustat | PAP: Placebo | LTTP: Eliglustat (Originally on Eliglustat) | LTTP: Eliglustat (Originally on Placebo)
Started | 20 | 20 | 0 | 0
Completed | 19 | 20 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: LTTP (Post-Week 39 up to Week 312)
Arm/Group | PAP: Eliglustat | PAP: Placebo | LTTP: Eliglustat (Originally on Eliglustat) | LTTP: Eliglustat (Originally on Placebo)
Started | 0 | 0 | 19 | 20
Completed | 0 | 0 | 12 | 15
Not Completed | 0 | 0 | 7 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Transitioned to commercial eliglustat | 0 | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) for PAP: included all participants who signed informed consent and received at least one dose of study drug (placebo or eliglustat).
Groups:
- PAP: Eliglustat: Eliglustat tartrate 50 mg capsule BID orally from Day 1 to Week 4, followed by eliglustat tartrate 50 mg or 100 mg capsule BID orally up to Week 39.
- Total: Total of all reporting groups
Arm/Group | PAP: Eliglustat | PAP: Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (11.55) | 32.1 (11.26) | 31.8 (11.26)
Gender [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 8 | 12 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Race: White | 19 | 20 | 39
  Race: Asian | 1 | 0 | 1
  Ethnicity: Not Hispanic or Latino | 18 | 20 | 38
  Ethnicity: Hispanic or Latino | 2 | 0 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated as ([weight in kg] divided by [height in cm multiplied by 0.01]^2).
  kilogram per square meter (kg/m^2) | 23.3 (2.74) | 23.4 (3.54) | 23.4 (3.13)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 64.8 (11.74) | 68.6 (17.17) | 66.7 (14.65)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.2 (9.91) | 170.0 (12.02) | 168.1 (11.05)

OUTCOME MEASURES:

1. Primary Outcome: PAP: Percent Change From Baseline in Spleen Volume (in Multiples of Normal [MN]) at Week 39 of the Primary Analysis Period With Eliglustat Tartrate Treatment as Compared to Placebo
Description: Percent change in spleen volume = ([spleen volume at Week 39 minus spleen volume at baseline] divided by [spleen volume at baseline]) multiplied by 100, where all volumes are in MN.
Time Frame: PAP Baseline (Day 1), Week 39
Population: FAS for PAP included all participants who signed informed consent and received at least one dose of study drug (placebo or eliglustat).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PAP: Eliglustat | PAP: Placebo
Number analyzed (Participants) | 20 | 20
percent change | -27.77 (2.37) | 2.26 (2.37)
Statistical Analysis 1: Comparison: PAP: Eliglustat vs PAP: Placebo; Analysis was performed using analysis of covariance (ANCOVA) model fitted with treatment and baseline spleen severity (low spleen severity: spleen volume less than or equal to [<=] 20 multiples of normal spleen volume, high spleen severity: spleen volume greater than [>] 20 multiples of normal spleen volume); Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -30.03, 95% CI 2-sided [-36.82 to -23.24], Standard Error of Mean 3.35

2. Secondary Outcome: PAP: Hemoglobin Level
Time Frame: PAP Baseline (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | PAP: Eliglustat | PAP: Placebo
Number analyzed (Participants) | 20 | 20
gram per deciliter (g/dL) | 12.05 (1.816) | 12.75 (1.629)

3. Secondary Outcome: PAP: Absolute Change From Baseline in Hemoglobin Level at Week 39
Description: Absolute change = hemoglobin level at Week 39 minus hemoglobin level at baseline.
Time Frame: PAP Baseline (Day 1), Week 39
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | PAP: Eliglustat | PAP: Placebo
Number analyzed (Participants) | 20 | 20
g/dL | 0.69 (0.23) | -0.54 (0.23)

4. Secondary Outcome: PAP: Percent Change From Baseline in Liver Volume (in MN) at Week 39
Description: Percent change in liver volume = ([liver volume at Week 39 minus liver volume at baseline] divided by [liver volume at baseline]) multiplied by 100, where all volumes are in MN.
Time Frame: PAP Baseline (Day 1), Week 39
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PAP: Eliglustat | PAP: Placebo
Number analyzed (Participants) | 20 | 20
percent change | -5.20 (1.64) | 1.44 (1.64)

5. Secondary Outcome: PAP: Percent Change From Baseline in Platelet Counts at Week 39
Description: Percent change in platelet count = ([platelet count at Week 39 minus platelet count at baseline] divided by [platelet count at baseline]) multiplied by 100.
Time Frame: PAP Baseline (Day 1), Week 39
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PAP: Eliglustat | PAP: Placebo
Number analyzed (Participants) | 20 | 20
percent change | 32.00 (5.95) | -9.06 (5.95)

6. Secondary Outcome: LTTP: Percent Change From Baseline in Spleen Volume (in MN) at Week 234
Description: Percent change in spleen volume = ([spleen volume at Week 234 minus spleen volume at baseline] divided by [spleen volume at baseline]) multiplied by 100, where all volumes are in MN. Baseline values for the original placebo participants refer to Day 1 of LTTP and baseline values for the original eliglustat participants refer to the Day 1 of PAP.
Time Frame: PAP Baseline for Eliglustat (Originally on Eliglustat) arm, LTTP Baseline for Eliglustat (Originally on Placebo) arm, Week 234
Population: Intent-to-treat (ITT) population for LTTP included all participants who received at least 1 dose of eliglustat in LTTP period. Number of participants analyzed= participants evaluable for this outcome measure and had available data for baseline and Week 234 spleen volume assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LTTP: Eliglustat (Originally on Eliglustat) | LTTP: Eliglustat (Originally on Placebo)
Number analyzed (Participants) | 7 | 6
percent change | -66.9 (8.45) | -64.0 (6.43)

7. Secondary Outcome: LTTP: Absolute Change From Baseline in Hemoglobin Level at Week 234
Description: Baseline values for the original placebo participants refer to Day 1 of LTTP and baseline values for the original eliglustat participants refer to the Day 1 of PAP.
Time Frame: as for outcome 6
Population: ITT population for LTTP included all participants who received at least 1 dose of eliglustat in LTTP period. Number of participants analyzed=participants evaluable for this outcome measure and had available data for baseline and Week 234 hemoglobin level assessment.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LTTP: Eliglustat (Originally on Eliglustat) | LTTP: Eliglustat (Originally on Placebo)
Number analyzed (Participants) | 7 | 5
g/dL | 1.1 (0.65) | 1.9 (1.88)

8. Secondary Outcome: LTTP: Percent Change From Baseline in Liver Volume (in MN) at Week 234
Description: Percent change in liver volume = ([liver volume at Week 234 minus liver volume at baseline] divided by [liver volume at baseline]) multiplied by 100, where all volumes are in MN. Baseline values for the original placebo participants refer to Day 1 of LTTP and baseline values for the original eliglustat participants refer to the Day 1 of PAP.
Time Frame: as for outcome 6
Population: ITT population for LTTP included all participants who received at least 1 dose of eliglustat in LTTP period. Number of participants analyzed=participants evaluable for this outcome measure and had available data for baseline and Week 234 liver volume assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LTTP: Eliglustat (Originally on Eliglustat) | LTTP: Eliglustat (Originally on Placebo)
Number analyzed (Participants) | 7 | 6
percent change | -24.3 (11.21) | -22.4 (10.77)

9. Secondary Outcome: LTTP: Percent Change From Baseline in Platelet Counts at Week 234
Description: Percent change in platelet count = ([platelet count at Week 234 minus platelet count at baseline] divided by [platelet count at baseline]) multiplied by 100. Baseline values for the original placebo participants refer to Day 1 of LTTP and baseline values for the original eliglustat participants refer to the Day 1 of PAP.
Time Frame: as for outcome 6
Population: ITT population for LTTP included all participants who received at least 1 dose of eliglustat in LTTP period. Number of participants analyzed=participants evaluable for this outcome measure and had available data for baseline and Week 234 platelet count assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LTTP: Eliglustat (Originally on Eliglustat) | LTTP: Eliglustat (Originally on Placebo)
Number analyzed (Participants) | 7 | 5
percent change | 77.3 (28.17) | 100.1 (80.69)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the signature of the Informed Consent Form through the follow-up period (30-37 days after the last visit, which was Week 312).
Description: Reported AEs are treatment-emergent that is AEs that developed/worsened during the 'on treatment period' (first dose of eliglustat to end of follow-up period).
Groups:
- Eliglustat: PAP: Eliglustat tartrate capsule 50 mg orally on Day 1 followed by eliglustat tartrate 50 mg capsule BID from Day 2 to Week 4, then either eliglustat tartrate 50 mg capsule BID(participants with Genz-99067 trough plasma concentration>=5 ng/mL) or eliglustat tartrate 100 mg capsule BID(participants with Genz-99067 trough plasma concentration<5 ng/mL), up to Week 39. PK assessment at Week 2 used for dose adjustment after Week 4. LTTP: Participants of the eliglustat arm in PAP who completed PAP were included in LTTP & received eliglustat tartrate capsule 50 mg BID orally from Day 1(post Week 39) until Week 43 followed by eliglustat tartrate 50 mg or 100 mg capsule BID up to Week 47, then eliglustat tartrate 50 mg or 100 mg or 150 mg capsule BID up to Week 312. Dose adjustments at Week 43 & Week 47 were based on Genz-99067 trough plasma concentrations(if trough plasma concentration<5 ng/mL: next higher dose administered;if>=5 ng/mL: same dose continued) at Week 41 & Week 45, respectively.
Arm/Group | Eliglustat | Placebo
Serious Adverse Events (participants affected / at risk) | 2/20 | 3/20
Other Adverse Events (participants affected / at risk) | 17/20 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat (N=20) | Placebo (N=20)
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat (N=20) | Placebo (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1
Palpitations (Cardiac disorders) | 0 | 3
Eye irritation (Eye disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 3 | 2
Toothache (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 3 | 1
Fatigue (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 2
Seasonal allergy (Immune system disorders) | 1 | 2
Bronchitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 3
Hordeolum (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 2
Otitis media (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 3 | 2
Tonsillitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Bone density decreased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 11 | 7
Migraine (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 2
Proteinuria (Renal and urinary disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.